CLINICAL TRIAL: NCT01824017
Title: Validation of RLIP76 Assay and Exploratory Study of RLIP76 Correlation Among Patients With Type 2 Diabetes and Metabolic Syndrome
Brief Title: Validation of an RLIP76 Assay in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12044
Record Dates: First submitted 2012-12-20; First posted 2013-04-04 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; metabolic syndrome; oxidative stress; GSH
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood Draw (Other): Data will be collected at patients' usual follow-up intervals for monitoring their metabolic conditions (i.e., T2D, hyperlipidemia, hypertriglyceridemia, etc.), which will be at 3 or 6 month intervals with a +/- 30 day window. Standard treatment surveillance measures such as hemoglobin A1c, LDL, and triglyceride levels will be performed as the standard of care for patients with MsY. Blood samples for these tests will be drawn while subjects are fasting
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw

SUMMARY:
The current proposal extends work done in mouse models evaluating the consistency of measuring RLIP76 in a clinical cohort (Aim 1) by using guidelines provided by the NIH for validating biomarkers. We will also proceed to estimate the effect size of a potential correlation of RLIP76 with standard MsY treatment measures such as hgbA1c, LDL, and triglyceride levels in a longitudinal prospective study ( Aim 2) that will follow a cohort of patients with MsY who seek care at the City of Hope Endocrine clinic over a 12 month period..

ELIGIBILITY:
Inclusion Criteria:

* Registered patient of City of Hope and followed in the Endocrine Clinic. Must have documentation of a diagnosis of diabetes identified by the problem list in the patient's electronic health record.
* Must demonstrate features of MsY by possessing any of the following characteristics and/or receiving treatment for diabetes, hyperlipidemia, and/or hypertriglyceridemia.

  * Central obesity: waist circumference ≥ 102 cm or 40 inches (male), ≥ 88 cm or 36 inches (female)
  * Dyslipidemia: TG ≥ 1.7 mmol/L (150 mg/dl)
  * Dyslipidemia: HDL-C < 40 mg/dL (male), < 50 mg/dL (female)
  * Blood pressure ≥ 130/85 mmHg
  * Fasting plasma glucose ≥ 6.1 mmol/L (110 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The consistency of an ELISA-based RLIP76 assay in the serum of human subjects with metabolic syndrome. | 12 months
  The investigators will perform 6 repeated measurements on first blood draws from patients with Type 2 diabetes who also have MsY. Sixty-seven percent (4 out of 6) of the quality controls must be within 15% of the mean of these measurements for us to consider the ELISA-based RLIP76 assay to be consistent

SECONDARY OUTCOMES:
Effect size of correlation of RLIP76 levels with treatment measures of metabolic syndrome such as hemoglobin A1c, LDL, and triglyceride levels. | 12 months
  The investigators will perform a longitudinal correlative study to evaluate the correlation of RLIP76 levels with changes in treatment measures of metabolic syndrome, such as hemoglobin A1c, LDL, and triglyceride levels. The results of this objective will be used to design a correlative study to determine the correlation of RLIP76 levels to the change in treatment measures of metabolic syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Raynald Samoa, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States